CLINICAL TRIAL: NCT06227910
Title: A Randomized, Double-Blind, Phase 3b Study to Evaluate the Short- and Long-Term Efficacy and Safety of Dual Targeted Therapy With Intravenous Vedolizumab and Oral Upadacitinib Compared With Intravenous Vedolizumab and Oral Placebo for Induction Followed by Intravenous Vedolizumab Monotherapy for Maintenance in the Treatment of Adults With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Vedolizumab With and Without Upadacitinib in Adults With Crohn's Disease
Acronym: VICTRIVA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-3043; 2023-509391-42-00 (EU CTIS Number: EU CT Number)
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind Induction Phase: Vedolizumab + Upadacitinib (Experimental): Participants will receive vedolizumab 300 mg intravenous (IV) infusion at Weeks 0, 2, 6 and 10 along with upadacitinib 45 mg, orally, once daily (QD) for 12 weeks.
  Interventions: Drug: Vedolizumab; Drug: Upadacitinib
- Double-blind Induction Phase: Vedolizumab + Placebo (Placebo Comparator): Participants will receive vedolizumab IV 300 mg infusion, at Weeks 0, 2, 6 and 10 along with upadacitinib matched placebo, orally, QD for 12 weeks.
  Interventions: Drug: Vedolizumab; Drug: Placebo
- Main Study Maintenance Phase: Vedolizumab Monotherapy (Experimental): Participants who achieve a CDAI reduction of >=70 points from baseline at Week 12 will receive vedolizumab 300 mg IV infusion (monotherapy), every 8 weeks (Q8W) starting at Week 14 to 52. The Q8W vedolizumab monotherapy may be escalated to Q4W at the investigator's discretion.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab IV infusion.
  Other Names: Entyvio; MLN0002; KYNTELES
Drug: Upadacitinib — Upadacitinib over-encapsulated tablets.
  Other Names: Rinvoq
  Arms: Double-blind Induction Phase: Vedolizumab + Upadacitinib
Drug: Placebo — Upadacitinib matched placebo capsules.
  Arms: Double-blind Induction Phase: Vedolizumab + Placebo

SUMMARY:
The main aim of this study is to learn whether vedolizumab and upadacitinib given together (also called dual targeted therapy or DTT) reduces bowel inflammation and ulcers in the bowel compared to vedolizumab only (also called monotherapy) in adults with moderately or severely active Crohn's Disease (CD) after 12 weeks of treatment. Other aims are to learn how safe and effective DTT is compared to monotherapy for these participants.

All participants will receive DTT (either vedolizumab and upadacitinib or vedolizumab and placebo) for 12 weeks. Participants responding to the treatment will then receive vedolizumab only (monotherapy) for an additional 40 weeks.

During the study, participants will visit their study clinic 15 times.

DETAILED DESCRIPTION:
The drug being tested in this study is vedolizumab. Vedolizumab is being tested to treat people with moderately to severely active CD. The study will look at the efficacy and safety of vedolizumab with and without upadacitinib. The study will enroll approximately 396 patients. Participants will be assigned in a 1:1 ratio to one of the two treatment groups in the 12-weeks Induction Phase:

* Induction Phase: Vedolizumab + Upadacitinib
* Induction Phase: Vedolizumab + Placebo

Participants who achieve a Crohn's disease activity index (CDAI) reduction of greater than or equal to (>=)70 points from baseline at Week 12 will enter the main study Maintenance Phase (40 weeks) of the study to receive vedolizumab monotherapy. Participants will be followed for a further 18-week safety follow-up period up to Week 70.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 70 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has a diagnosis of CD established at least 3 months before screening by clinical and endoscopic evidence and corroborated by a histopathology report.
2. The participant has a confirmed diagnosis of moderately to severely active CD as assessed by CDAI of 220-450.
3. The participant has evidence of mucosal inflammation based on the SES-CD: SES-CD score (excluding the presence of narrowing component) of >=6 (or >=4 for participants with isolated ileal disease), as confirmed by a central reader.
4. The participant has demonstrated an inadequate response to, loss of response to, or intolerance to corticosteroids, immunomodulators, or biologic therapy.

Exclusion Criteria:

1. The participant has a current diagnosis of ulcerative colitis or indeterminate colitis.
2. The participant has infection(s) requiring treatment with IV anti-infectives within 30 days prior to baseline or oral/intramuscular anti-infectives within 14 days prior to baseline.
3. The participant has evidence of an active infection during the screening period, or clinically significant infection within 30 days prior to screening, or ongoing chronic infection.
4. The participant has a history of recurrent or disseminated (including a single episode) herpes zoster, or disseminated (including a single episode) herpes simplex.
5. The participant has any of the following ongoing known complications of CD: abscess (abdominal or peri-anal); symptomatic bowel strictures; 2 entire missing segments of the following 5 segments: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum; fulminant colitis; toxic megacolon; or any other manifestation that might require surgery while enrolled in the study.
6. The participant has an ostomy or ileoanal pouch.
7. The participant has severe renal impairment, defined as an estimated glomerular filtration rate of <30 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2).
8. The participant has severe (Child-Pugh C) hepatic impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission Based on the CDAI at Week 12 | Week 12
  Clinical remission is defined as a CDAI score of <150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit, and body weight. CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of Participants Exhibiting an Endoscopic Response Based on Simple Endoscopic Score for CD (SES-CD) at Week 12 | Week 12
  Endoscopic response per SES-CD is assessed as proportion of participants achieving decrease in SES CD >50% from baseline (for participants with isolated ileal disease,SES-CD <=4 or <=2-point reduction from baseline) read centrally. SES-CD evaluates 4 endoscopic variables (ulcer size,percentage of ulcerated and affected surface area,presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy (ileum,right,transverse,and left colon,rectum). Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of the scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. Overall SES-CD score ranges from 0 to 56 and is sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving 2-item Patient-reported Outcome Measure (PRO2) Based Clinical Remission at Week 12 | Week 12
  Clinical remission based on PRO2 is defined as 7-day average of very soft or liquid stool frequency (SF) <=2.8, 7-day average of abdominal pain (AP) score <=1.0, and neither worse than baseline. The PRO2 is comprised of the stool frequency and abdominal pain components of the CDAI.
Percentage of Participants Achieving Endoscopic Remission Based on SES-CD at Week 12 | Week 12
  Endoscopic remission as per SES-CD is defined as an SES-CD score of ≤4 with no mucosal ulceration in the colon or ileum as assessed by centrally read video ileocolonoscopy. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of surface area (SA) that is ulcerated, percentage of SA affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.
Percentage of Participants Exhibiting Corticosteroid-free Clinical Remission in Participants who Were Taking Corticosteroids at Baseline Based on the CDAI at Week 12 | Week 12
  Percentage of participants using oral corticosteroids at Baseline who have discontinued corticosteroids and are in clinical remission per CDAI at Week 12 will be reported. Clinical remission is defined as a CDAI score of <150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit, and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of Participants Exhibiting a Clinical Response Based on the CDAI at Week 12 | Week 12
  Clinical response is defined as >=100-point decrease from Baseline in CDAI score. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit, and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of Participants Achieving Clinical Remission Based on the CDAI at Week 52 | Week 52
  Clinical remission is defined as a CDAI score of <150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit, and body weight. CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of Participants Exhibiting an Endoscopic Response Based on SES-CD at Week 52 | Week 52
  Endoscopic response per SES-CD is assessed as proportion of participants achieving decrease in SES CD >50% from baseline (for participants with isolated ileal disease,SES-CD <=4 or <=2-point reduction from baseline) read centrally. SES-CD evaluates 4 endoscopic variables (ulcer size,percentage of ulcerated and affected surface area,presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy (ileum,right,transverse,and left colon,and rectum). Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. Overall SES-CD score ranges from 0 to 56 and is sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.
Percentage of Participants Achieving 2-item PRO2 Based Clinical Remission at Week 52 | Week 52
  Clinical remission based on PRO2 is defined as 7-day average of very soft or liquid stool frequency (SF) <=2.8, 7-day average of abdominal pain (AP) score <=1.0, and neither worse than baseline. The PRO2 is comprised of the stool frequency and abdominal pain components of the CDAI.
Percentage of Participants Achieving Endoscopic Remission Based on SES-CD at Week 52 | Week 52
  Endoscopic remission as per SES-CD is defined as an SES-CD score of <=4 with no mucosal ulceration in the colon or ileum as assessed by centrally read video ileocolonoscopy. SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of surface area (SA) that is ulcerated, percentage of SA affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy. Each variable is coded from 0 to 3 based on severity, where 0 is none or not severe and 3 is most severe case, with sum of scores for each variable ranging from 0 to 15, except for presence of narrowing. Presence of narrowing ranges from 0 to 11 since a severity of 3 represents a narrowing which a colonoscope cannot be passed and, thus, can only be observed once among the bowel segments. The overall SES-CD score ranges from 0 to 56 and is sum of 4 variables across 5 bowel segments. Higher scores indicate more severe disease.
Percentage of Participants Exhibiting Corticosteroid-free Clinical Remission in Participants who Were Taking Corticosteroids at Baseline Based on the CDAI at Week 52 | Week 52
  Percentage of participants using oral corticosteroids at Baseline who have discontinued corticosteroids and are in clinical remission at Week 52 per CDAI will be reported. Clinical remission is defined as a CDAI score of <150 points. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit, and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of Participants Exhibiting a Clinical Response Based on the CDAI at Week 52 | Week 52
  Clinical response is defined as >=100-point decrease from Baseline in CDAI score. CDAI assesses CD based on clinical signs such as number of liquid or very soft stools, abdominal pain, general wellbeing, extra-intestinal manifestations of CD, antidiarrheal use, presence of abdominal mass, hematocrit, and body weight. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (138):
- United States (19):
  - UCSD Medical Center, La Jolla, California
  - Keck Medicine Of USC - USC Healthcare Center 1, Los Angeles, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - GI PROS, Inc., Naples, Florida
  - Orlando Health Ambulatory Care Center, Orlando, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Indiana University (IU) Health University Hospital, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Mount Sinai Hospital - The Susan and Leonard Feinstein Inflammatory Bowel Disease (IBD) Clinical Center, New York, New York
  - Columbia University Medical Center, New York-Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital Northwell Health, New York, New York
  - Gastroenterology Associates, Greenville, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Medical College of Wisconsin Cancer Center - Froedtert Hospital, Milwaukee, Wisconsin
- Austria (5):
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Medizinische Universitaet Wien - Allgemeines Krankenhaus der Stadt Wien (AKH) - Universitaetsklinik fuer Innere Medizin III, Vienna, Vienna
  - Johannes Kepler Universitat Linz (JKU), Linz
  - Landeskrankenhaus Salzburg, Innere Medizin I, Labor im Erdgeschoss, Salzburg
  - Krankenhaus der Barmherzigen Brueder Wien, Vienna
- Belgium (5):
  - Hopital Universitaire de Bruxelles/ Academisch Ziekenhuis Brussel, Brussels, Anderlecht
  - Imelda GI Clinical Research Center, Bonheiden
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospitals Leuven, Leuven
  - Centre Hospitalier Chretien MontLegia, Liège
- Brazil (7):
  - Hospital Universitario Cajuru, Curitiba, Paraná
  - Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Centro de Estudos Clinico do Interior Paulista - CECIP, Jaú, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - Universidade Federal do Rio de Janeiro (UFRJ)-Hospital Universitario Clementino Fraga Filho (HUCFF), Rio de Janeiro
  - Hospital das Clinicas of the University of Sao Paulo (Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo (HC/FMUSP)), São Paulo
  - Unidade de Pesquisa Clinica UPC Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, São Paulo
- Canada (9):
  - Heritage Medical Research Clinic - University Of Calgary, Calgary, Alberta
  - University of Manitoba-Winnipeg Regional Health Authority-Health Sciences Centre, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Barrie GI Associates, Barrie, Ontario
  - McMaster University - Farncombe Family Digestive Health Research Institute (FFDHRI), Hamilton, Ontario
  - Taunton Surgical Centre-Oshawa Clinic, Oshawa, Ontario
  - Toronto Immune and Digestive Health Institute (TIDHI), Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Croatia (3):
  - Poliklinika Borzan d.o.o., Osijek
  - Clinical Hospital Center Rijeka, Rijeka
  - University Hospital Centre Sestre Milosrdnice, Zagreb
- Czechia (4):
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - IBD Clinical and Research centre, Prague
- Denmark (2):
  - Aalborg Hospital, Aalborg
  - Hvidovre Hospital Medicinsk Gastroenterologisk Afdeling, Hvidovre
- France (8):
  - CHU d'Amiens-Picardie - Hopital SUD, Amiens
  - Hopital Huriez - CHRU de Lille, Lille
  - Chu - Hopital Nord, Marseille
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hopital Hotel Dieu, Nantes
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut-Leveque, Pessac
  - CHU St Etienne Hopital Nord, Saint-Etienne
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital Rangueil, Toulouse
  - Centre Hospitalier Regional Universitaire de Nancy, Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Krankenhaus Waldfriede e.V., Berlin
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Studiengesellschaft BSF, Halle
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein, UKSH-Campus Kiel, Kiel
  - St. Marien- und St. Annastiftskrankenhaus, Ludwigshafen
  - Universitaetsklinikum Mannheim (Umm) - Ii Medizinische Klinik, Mannheim
- Greece (3):
  - University of Athens School of Medicine, Alexandra General Hospital, Athens, Attica
  - Metaxa Cancer Hospital, Piraeus, Attica
  - University Hospital of Heraklion, Heraklion, Crete
- Hungary (3):
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Semmelweis Egyetem, Budapest
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Szent-Gyorgyi Albert Klinikai Kozpont, I.Sz. Belogyaszati Klinika, Szeged
- Ireland (3):
  - Adelaide, Meath and National Children's Hospital, Dublin
  - University College Dublin (UCD) - St. Vincent's University Hospital (SVUH), Dublin
  - Beaumont Hospital, Dublin
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus (RHCC), Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Beilinson Campus (Beilinson and Hasharon Hospital), Petah Tikva
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Ospedale San Raffaele (HSR) Instituto Scientifico Universitario San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Federico II di Napoli, Naples
  - A. Gemelli University Hospital, Catholic University of the Sacred Heart, Roma
  - Humanitas Clinical And Research Institute, Rozzano
  - Fondazione IRCSS Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - AO Ordine Mauriziano di Torino, Torino
- Netherlands (4):
  - Amsterdam UMC Research BV, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Elisabeth TweeSteden Ziekenhuis (ETZ), Tilburg
- Norway (4):
  - Vestre Viken HF - Baerum Sykehus, Drammen, Gjettum
  - Haukeland Universitetssjukehus (Haukeland University Hospital), Bergen
  - Akershus University Hospital, Lorenskog
  - Oslo Universitetssykehus HF, Ulleval, Oslo
- Poland (5):
  - Oddzial Kliniczny Gastroenterologii Ogolnej i Onkologicznej SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Im. H. Swiecickiego Um, Poznan
  - H-T. Centrum Medyczne Sp. z o.o. Sp.k., Tychy
  - Panstwowy Instytut Medyczny MSWiA, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Portugal (3):
  - Unidade Local de Saude Coimbra, Coimbra
  - Centro Hospitalar de Lisboa ocidental (CHLO), Hospital Egas Moniz, Lisbon
  - Centro Hospitalar Universitario Lisboa Norte EPE, Lisbon
- University Clinical Centre - Ljubljana, Ljubljana, Slovenia
- South Korea (8):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea, Daejeon St.Mary's Hospital, Daejeon
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - The Catholic University Of Korea, St. Vincent's Hospital, Suwon
- Spain (6):
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari Son Espases, Palma
  - Complejo Hospitalario de Navarra (CHN), Pamplona
  - Complejo Hospitalario Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Universitari I Politecnic La Fe, Valencia
- Sweden (4):
  - Universitetssjukhuset i Linkoping, Endokrin- och magtarmmedicinska Kliniken (EM-Kliniken), Linköping
  - Ersta sjukhus, Stockholm
  - Karolinska Universitetssjukhuset - Hjartkliniken i Solna - Karolinska University Hospital, Stockholm
  - Danderyds Sjukhus AB, Stockholm
- Switzerland (4):
  - University Hospital Basel, Basel
  - University Hospital Bern (Inselspital), Bern
  - Zentrum fur Gastroenterologie, Zurich
  - Universitatsspital Zurich, Zurich
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Defense Medical Center (NDMC) (Tri-Service General Hospital (TSGH)) - Neihu, Taipei
  - Chang Gung Memorial Foundation Linkou Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (4):
  - St Thomas' Hospital - Guy's & St Thomas' NHS Foundation Trust, London, England
  - The Royal London Hospital - Barts Health NHS Trust, London, Greater London
  - Western General Hospital, Edinburgh, Lothian
  - Queen Elizabeth University Hospital - NHS Greater Glasgow & Clyde - South Glasgow University Hospital Division, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Danese S, Sands BE, Feagan BG, Jairath V, Panaccione R, Peyrin-Biroulet L, Irving PM, Schreiber S, Dotan I, Ferrante M, D'Haens GR, Jones S, Freire M, Lindner D, Adsul S, Oberai P, Colombel JF. Design and rationale for the VICTRIVA study: A randomized, double-blind, phase 3b study of vedolizumab in combination with upadacitinib in Crohn's disease. Contemp Clin Trials Commun. 2025 Nov 24;48:101574. doi: 10.1016/j.conctc.2025.101574. eCollection 2025 Dec. PMID 41403476
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/cffb4e6c789e4ac4?idFilter=%5B%22Vedolizumab-3043%22%5D